CLINICAL TRIAL: NCT00763087
Title: Effect of Weight-Bearing Exercise on People With Diabetes and Neuropathic Feet
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 06-0953
Record Dates: First submitted 2008-09-26; First posted 2008-09-30 (Estimated); Last update posted 2017-11-07 (Actual); Status verified 2017-11

CONDITIONS: Diabetes Mellitus; Peripheral Neuropathy
Keywords: diabetes mellitus; peripheral neuropathy; exercise
MeSH Terms: conditions — Diabetes Mellitus; Peripheral Nervous System Diseases; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- nonweightbearing exercise (Active Comparator)
  Interventions: Behavioral: nonweightbearing exercise
- nonexercising control (Placebo Comparator)
  Interventions: Behavioral: nonexercising control
- weightbearing exercise (Experimental)
  Interventions: Behavioral: weightbearing exercise

INTERVENTIONS:
Behavioral: weightbearing exercise — All subjects in the exercise group will participate, as able, in 3 supervised 1 hour exercise sessions per week for the first month and 2 supervised and 1 unsupervised exercise session per week for the remaining 2 months. Subjects in each exercise group will be seen on alternating times to avoid cross contamination of treatment intervention. Walking intensity for all subjects will be applied with the intent to exceed their routine physical stress level, and therefore incur positive adaptations to physical stress, but not exceed their threshold for injury.
  Arms: weightbearing exercise
Behavioral: nonweightbearing exercise — All subjects in the 2 exercise groups will participate, as able, in 3 supervised 1 hour exercise sessions per week for the first month and 2 supervised and 1 unsupervised exercise session per week for the remaining 2 months. Subjects in each exercise group will be seen on alternating times to avoid cross contamination of treatment intervention. Biking intensity for all subjects will be applied with the intent to exceed their routine physical stress level, and therefore incur positive adaptations to physical stress, but not exceed their threshold for injury.
  Arms: nonweightbearing exercise
Behavioral: nonexercising control — All subjects will be instructed, verbally and with written documents, regarding appropriate foot and skin care twice per month.
  Arms: nonexercising control

SUMMARY:
The purpose of this study is to determine if people with Diabetes Mellitus and peripheral neuropathy can increase their activity (i.e. walking or stationary biking) and leg strength without having an increase in foot problems compared to a group of people with diabetes and peripheral neuropathy that do no exercise.

Our hypothesis is that the weight-bearing exercise group will achieve greater increases in weight-bearing activity (i.e., increased steps/day and cumulative load) and leg strength compared to the non-weight bearing exercise group and the non-exercising control group; and there will be no clinically meaningful difference in incidence or indicators of foot lesions between groups.

DETAILED DESCRIPTION:
People with diabetes and peripheral neuropathy (DM+PN) have substantial lower extremity impairments, functional limitations and disability. In addition to muscle weakness and poor balance, they also are at high risk for foot ulcerations, especially if they have a history of ulceration. Although there is a large and growing body of knowledge about the effect of exercise on people with DM, there is little evidence about the effect of exercise in people with DM+PN. Exercise is an important treatment component to help control the complications of DM. The American Diabetes Association (ADA), and the American College of Sports Medicine (ACSM)4 recommend that adults with DM participate in at least 30 minutes a day of moderate-intensity physical activity that is consistent with a brisk walk. The ADA and ACSM, however, discourage weight-bearing exercise for people with DM+PN due to risk of exercise-induced foot injury. No data support this guideline to restrict those with DM+PN from weight-bearing activity, and in fact, some evidence suggests that those with DM+PN who are most active are least likely to develop skin breakdown. The Primary Goal of this proposal is to conduct a pilot randomized prospective controlled clinical trial to determine if people with DM+PN can benefit from a progressive weight-bearing exercise program to improve impairments, functional limitations, disability, and pathophysiology without an increase in skin breakdown or foot lesions. The benefits of a weight bearing program will be compared to the benefits of a non weight bearing exercise program and to a non-exercising control group. The results of this study also will help to determine if neuropathic skin and muscle can adapt to increasing physical stress levels without injury which could have important implications for weight-bearing and exercise guidelines for people with DM+PN.

A. SPECIFIC AIMS

Aim 1. Determine the effect of a weight-bearing exercise program compared to a non-weight bearing exercise program and to a non-exercising control group on indicators of impairments, functional limitations, disability, and pathophysiology in patients with DM+PN.

1. Measures of Impairment: Ankle joint range of motion, ankle plantar flexor and dorsiflexor muscle strength (peak torque), muscle volume (magnetic resonance imaging), and standing balance.

   H1: Both exercise groups will show an improvement in ankle joint range of motion and ankle plantar flexor / dorsiflexor muscle strength / volume compared to the non-exercising control group, but only the weight-bearing exercise group will show an improvement in standing balance because of exposure to challenging weight-bearing activities.
2. Measures of Functional Limitations: Physical Performance Test, Foot & Ankle Ability Measure.

   H2: Both exercise groups will show improvement in the Physical Performance Test and Foot & Ankle Ability Measure compared to the non-exercising control group, and the weight-bearing exercise group will show greater improvements than the non-weight bearing exercise group because of improved balance and exposure to challenging weight-bearing activities.
3. Measures of Disability / Participation: Diabetes Symptom Checklist, Beck Depression Inventory.

   H3: Both exercise groups will show improved measures of disability compared to the non-exercising control group, and the weight-bearing exercise group will show greater improvements than the non-weight bearing exercise group because of improved ability to participate in community activities which require weight-bearing and walking ability.
4. Measures of Pathophysiology: HbA1c, serum lipids, DXA (body composition), and body mass index.

H4: Both exercise groups will show modest but statistically significant improvements compared to the non-exercising control group in the above measures of pathophysiology.

Aim 2: Determine the effect of weight-bearing exercise program and non-weight bearing exercise program compared to a control group on 1) daily step count (steps/day), 2) an estimate of cumulative load (step count * plantar pressure integral), 3) unilateral increase in surface foot temperature, and 4) incidence of foot lesions (digital photograph).

H5: The weight-bearing exercise group will achieve greater increases in weight-bearing activity (i.e., increased steps/day and cumulative load) compared to the non-weight bearing exercise group and the non-exercising control group; and there will be no clinically meaningful difference in incidence or indicators of foot lesions between groups.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 or Type 2 DM and PN
* biothesiometer > 25mV and
* unable to sense the 5.07 Semmes Weinstein monofilament on at least one spot on the plantar foot
* Relatively sedentary
* step count of 2-9,000 steps per day
* exercising less than 3 times per week (<20 min/session).
* Have the approval of his/her primary care physician to participate in the study.

Exclusion Criteria:

* Subjects who weigh greater than 300 pounds (DXA scanner's weight limit).
* A history of severe foot deformity, such as Charcot neuroarthropathy or partial foot amputation that would require custom therapeutic footwear.
* Any co-morbidity or medication that would interfere with ability to exercise according to ADA and ACSM guidelines.
* People with severe depression as determined by the Beck Depression Inventory II with a score of 29 or greater.
* People who are physically incapable of tolerating one hour of activity.
* Women of child bearing age due to risk of exposure from radiation in DXA testing.

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2008-09; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
daily step count | 3 months

SECONDARY OUTCOMES:
skin breakdown | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Mueller, PT, PhD, Principal Investigator — Washington University in St. Louis, Program in Physical Therapy
Locations (1):
- Program in Physical Therapy, Washington University in St. Louis, St Louis, Missouri, United States